CLINICAL TRIAL: NCT01721473
Title: Nicotinic Acetylcholine Receptor Density and Veteran Cigarette Smokers
Brief Title: Brain Nicotine Receptor Density in Veteran Smokers
Acronym: BNRDVS
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: NURA-02-11S
Record Dates: First submitted 2012-10-29; First posted 2012-11-05 (Estimated); Results first posted 2019-10-07 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: Positron Emission Tomography
Keywords: Tobacco; Positron Emission Tomography; Marijuana; Caffeine; Menthol
MeSH Terms: conditions — Marijuana Abuse | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — None retained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- cigarette smokers with heavy marijuana use: With heavy marijuana use
  Interventions: Other: positron emission tomography scan
- cigarette smokers with heavy caffeine use: with heavy caffeine use
  Interventions: Other: positron emission tomography scan
- cigarette smokers w/o heavy caffeine and marijuana use: cigarette smokers without the heavy use of marijuana or caffeine
  Interventions: Other: positron emission tomography scan
- non-smokers: not a regular cigarette user
  Interventions: Other: positron emission tomography scan
- cigarette smokers with non-menthol cigarette preference: non-menthol cigarette preference
  Interventions: Other: positron emission tomography scan
- cigarette smokers with menthol cigarette preference: menthol cigarette preference
  Interventions: Other: positron emission tomography scan

INTERVENTIONS:
Other: positron emission tomography scan — 2-FA positron emission tomography scan

SUMMARY:
Cigarette smoking is more prevalent among Veterans (27%) than the general U.S. population (21%). Smoking is common among people who use marijuana or caffeine heavily, and the use of menthol cigarettes is becoming increasingly common, affecting approximately 9% of the Veteran population. Recent research by the group and others indicates that heavy marijuana or caffeine use, or the use of predominantly menthol cigarettes, can alter brain nicotinic acetylcholine receptor (nAChR) densities. For the proposed study, brain imaging with PET scanning will be used to determine nicotine receptor densities in Veteran cigarette smokers with and without heavy marijuana or caffeine use, and in menthol and non-menthol Veteran smokers. Results of the proposed research may have implications for improving treatments for Veterans who smoke cigarettes and who have specific drug use co-morbidities or who use menthol cigarettes.

DETAILED DESCRIPTION:
Despite improvements in tobacco control, the prevalence of Tobacco Dependence (TD) remains high at 27% among Veterans and 21% among the general U.S. population (~46 million U.S. adults). Both co-morbid substance use and menthol cigarette preference are important issues contributing to greater severity of TD. Among smokers, a lifetime history of substance use/dependence is common and approximately 33% of all smokers use primarily menthol cigarettes, meaning that roughly 9% of Veterans smoke menthol. In addition to menthol cigarette usage being prevalent among Veterans, this problem is likely to worsen over time, because recent military deployments increase the chances of smoking initiation and marketing of menthol cigarettes is aimed at roughly the age group that comprises the active military.

For substance use/dependence, marijuana (MJ) users are five times more likely than non-MJ users to smoke tobacco cigarettes, and regular caffeine users are twice as likely as non-caffeine users to smoke cigarettes. Cigarette smoking contributes greatly to morbidity and mortality among patients with drug (and alcohol) dependencies, making it vital to understand better the complex relationship between drug/alcohol dependence and brain nicotine receptor densities in cigarette smokers.

Based on prior literature and pilot data collected during the previous Merit Review period, the primary hypotheses for the proposed research are that: 1) Participants who are heavy MJ users will have higher 4 2* nAChR densities in the thalami (and other brain regions) than participants who are not heavy MJ users, 2) Participants who are daily heavy caffeine users will have lower 4 2* nAChR densities in the thalami (and other regions) than participants who are not heavy daily caffeine users, 3) Densities of 4 2* nAChRs in the thalami (and other brain regions of interest) will be higher in menthol than non-menthol cigarette smokers, and 4) lesser severity of 4 2* nAChR up-regulation at baseline (along with clinical factors such as lesser severity of nicotine dependence) will be associated with better treatment outcomes in a standard smoking cessation program, including an improved likelihood of quitting and/or decreasing smoking.

To test these hypotheses, cigarette smokers will be recruited through flyers posted at the VA Greater Los Angeles Healthcare System in areas where smokers are likely to be present. Participants will undergo the following sequence of procedures: (1) telephone/in-person screening, (2) a bolus-plus-continuous-infusion 2-FA positron emission tomography (PET) scanning session, (3) a structural magnetic resonance imaging scan within one week of the initial PET session, and (4) referral to a standard 12-week smoking cessation program. Rating scales for the determination of smoking-related symptoms will be collected before and during the PET scanning procedure. Smoking status and measures of nicotine exposure and metabolism will be collected during the study using participant reports, exhaled carbon monoxide (CO) levels, urine cotinine levels, and plasma nicotine, cotinine, and 3'-hydroxycotinine levels.

ELIGIBILITY:
Inclusion Criteria:

* Must be a Veteran cigarette smoker, living within commuting distance of the VA San Diego Healthcare System
* Healthy adult Veterans (18 to 65 years old) who are tobacco dependent cigarette smokers (10 to 40 cigarettes per day) meeting criteria for Nicotine Dependence as defined by DSM-IV criteria109 and who want to quit smoking.
* Heavy marijuana or caffeine use (defined as using the equivalent of > 2 marijuana cigarettes per week or the use of at least 3 coffee cup equivalents per day) for at least the past 6 months or no heavy drug/alcohol use.
* Ability to read, write, and give voluntary informed consent.
* An exhaled CO > 8 ppm during the study screening visit to verify smoking status.

Exclusion Criteria:

* Any Axis I diagnosis (including mood, anxiety, and psychotic disorders) other than Nicotine, Marijuana, or Caffeine Dependence within the past 1 year.
* A current diagnosis (within the past month) of other substance abuse/dependence diagnoses (such as cocaine, amphetamine, or opiates). (Length of abstinence will be verified through participant interview and a chart review at the initial study visit, which typically includes information about substance abuse treatment history and objective verification with breathalyzer and/or urine toxicology screens). Occasional drug/alcohol use not meeting criteria for abuse/dependence will not be exclusionary.
* Any current medication or any history of a medical condition that might affect the central nervous system at the time of scanning (e.g., current treatment with a psychotropic medication, or history of severe head trauma with loss of consciousness, epilepsy, or other neurological diseases).
* The combination of both heavy marijuana and caffeine use.
* Unstable cardiovascular disease, severe liver disease, or renal insufficiency, which might make tolerating study procedures difficult. Routine history and physical examination will be performed at the initial screening visit to insure that participants meet study criteria (Section D4).
* Pregnancy (urine pregnancy tests will be obtained on all women of childbearing potential) due to the theoretical risk of radiation exposure to the fetus.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans who are cigarette smokers (10 to 40 cigarettes per day) who either use significant amounts of caffeine or marijuana (or who have little or no such use).
Sampling Method: Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur L Brody, MD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (2):
- United States (2):
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Potenza MN, Brody AL. Commentary on Boileau et al. (2013): Distinguishing D2/D3 dopaminergic contributions to addictions. Addiction. 2013 May;108(5):964-5. doi: 10.1111/add.12119. No abstract available. PMID 23587083
- [Background] Jasinska AJ, Zorick T, Brody AL, Stein EA. Dual role of nicotine in addiction and cognition: a review of neuroimaging studies in humans. Neuropharmacology. 2014 Sep;84:111-22. doi: 10.1016/j.neuropharm.2013.02.015. Epub 2013 Mar 6. PMID 23474015
- [Background] Brody AL, Mukhin AG, Stephanie Shulenberger, Mamoun MS, Kozman M, Phuong J, Neary M, Luu T, Mandelkern MA. Treatment for tobacco dependence: effect on brain nicotinic acetylcholine receptor density. Neuropsychopharmacology. 2013 Jul;38(8):1548-56. doi: 10.1038/npp.2013.53. Epub 2013 Feb 21. PMID 23429692
- [Background] Jarcho JM, Feier NA, Bert A, Labus JA, Lee M, Stains J, Ebrat B, Groman SM, Tillisch K, Brody AL, London ED, Mandelkern MA, Mayer EA. Diminished neurokinin-1 receptor availability in patients with two forms of chronic visceral pain. Pain. 2013 Jul;154(7):987-96. doi: 10.1016/j.pain.2013.02.026. Epub 2013 Mar 5. PMID 23582152
- [Background] Storage S, Mandelkern MA, Phuong J, Kozman M, Neary MK, Brody AL. A positive relationship between harm avoidance and brain nicotinic acetylcholine receptor availability. Psychiatry Res. 2013 Dec 30;214(3):415-21. doi: 10.1016/j.pscychresns.2013.07.010. Epub 2013 Oct 19. PMID 24148908
- [Background] Xu J, Fregni F, Brody AL, Rahman AS. Transcranial direct current stimulation reduces negative affect but not cigarette craving in overnight abstinent smokers. Front Psychiatry. 2013 Sep 20;4:112. doi: 10.3389/fpsyt.2013.00112. eCollection 2013. PMID 24065930
- [Background] Le Foll B, Guranda M, Wilson AA, Houle S, Rusjan PM, Wing VC, Zawertailo L, Busto U, Selby P, Brody AL, George TP, Boileau I. Elevation of dopamine induced by cigarette smoking: novel insights from a [11C]-+-PHNO PET study in humans. Neuropsychopharmacology. 2014 Jan;39(2):415-24. doi: 10.1038/npp.2013.209. Epub 2013 Aug 19. PMID 23954846
- [Background] Zanchi D, Brody AL, Montandon ML, Kopel R, Emmert K, Preti MG, Van De Ville D, Haller S. Cigarette smoking leads to persistent and dose-dependent alterations of brain activity and connectivity in anterior insula and anterior cingulate. Addict Biol. 2015 Nov;20(6):1033-41. doi: 10.1111/adb.12292. Epub 2015 Aug 25. PMID 26303184
- [Background] Brody AL, Zorick T, Hubert R, Hellemann GS, Balali S, Kawasaki SS, Garcia LY, Enoki R, Abraham P, Young P, McCreary C. Combination Extended Smoking Cessation Treatment Plus Home Visits for Smokers With Schizophrenia: A Randomized Controlled Trial. Nicotine Tob Res. 2017 Jan;19(1):68-76. doi: 10.1093/ntr/ntw190. Epub 2016 Aug 3. PMID 27613888
- [Background] Xie J, Douglas PK, Wu YN, Brody AL, Anderson AE. Decoding the encoding of functional brain networks: An fMRI classification comparison of non-negative matrix factorization (NMF), independent component analysis (ICA), and sparse coding algorithms. J Neurosci Methods. 2017 Apr 15;282:81-94. doi: 10.1016/j.jneumeth.2017.03.008. Epub 2017 Mar 18. PMID 28322859
- [Result] Brody AL, Mukhin AG, La Charite J, Ta K, Farahi J, Sugar CA, Mamoun MS, Vellios E, Archie M, Kozman M, Phuong J, Arlorio F, Mandelkern MA. Up-regulation of nicotinic acetylcholine receptors in menthol cigarette smokers. Int J Neuropsychopharmacol. 2013 Jun;16(5):957-66. doi: 10.1017/S1461145712001022. Epub 2012 Nov 21. PMID 23171716
- [Result] Brody AL, Mukhin AG, Mamoun MS, Luu T, Neary M, Liang L, Shieh J, Sugar CA, Rose JE, Mandelkern MA. Brain nicotinic acetylcholine receptor availability and response to smoking cessation treatment: a randomized trial. JAMA Psychiatry. 2014 Jul 1;71(7):797-805. doi: 10.1001/jamapsychiatry.2014.138. PMID 24850280
- [Result] Zorick T, Mandelkern MA, Brody AL. A naturalistic study of the association between antidepressant treatment and outcome of smoking cessation treatment. J Clin Psychiatry. 2014 Dec;75(12):e1433-8. doi: 10.4088/JCP.14m09012. PMID 25551240
- [Result] Brody AL, McClernon FJ. Prediction of smoking cessation with treatment: the emerging contribution of brain imaging research. Neuropsychopharmacology. 2015 May;40(6):1309-10. doi: 10.1038/npp.2015.31. No abstract available. PMID 25868069
- [Result] Dubroff JG, Doot RK, Falcone M, Schnoll RA, Ray R, Tyndale RF, Brody AL, Hou C, Schmitz A, Lerman C. Decreased Nicotinic Receptor Availability in Smokers with Slow Rates of Nicotine Metabolism. J Nucl Med. 2015 Nov;56(11):1724-9. doi: 10.2967/jnumed.115.155002. Epub 2015 Aug 13. PMID 26272810
- [Result] Brody AL, Hubert R, Mamoun MS, Enoki R, Garcia LY, Abraham P, Young P, Mandelkern MA. Nicotinic acetylcholine receptor availability in cigarette smokers: effect of heavy caffeine or marijuana use. Psychopharmacology (Berl). 2016 Sep;233(17):3249-57. doi: 10.1007/s00213-016-4367-x. Epub 2016 Jul 1. PMID 27370018
- [Result] Brody AL, Hubert R, Enoki R, Garcia LY, Mamoun MS, Okita K, London ED, Nurmi EL, Seaman LC, Mandelkern MA. Effect of Cigarette Smoking on a Marker for Neuroinflammation: A [11C]DAA1106 Positron Emission Tomography Study. Neuropsychopharmacology. 2017 Jul;42(8):1630-1639. doi: 10.1038/npp.2017.48. Epub 2017 Mar 6. PMID 28262740

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-smokers: People who did not smoke or use heavy caffeine or marijuana
- Menthol Smokers: People who smoke menthol cigarettes.
- Non-menthol Smokers: People who smoke non-menthol cigarettes
- Smokers Without Comorbidities: People who smoke without heavy caffeine or marijuana use.
- Smokers With Caffeine: People who smoke and have heavy caffeine use.
- Smokers With Marijuana: People who smoke and heavily use marijuana.
Period: Overall Study
Arm/Group | Non-smokers | Menthol Smokers | Non-menthol Smokers | Smokers Without Comorbidities | Smokers With Caffeine | Smokers With Marijuana
Started | 47 | 22 | 41 | 34 | 22 | 18
Completed | 47 | 22 | 41 | 34 | 22 | 18
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Non-smokers: People who did not smoke.
- Smokers Methol: People who smoke menthol cigarettes.
- Smokers Non Menthol: People who smoke non menthol cigarettes.
- Smokers Without Comorbidities: People who smoke but do not have heavy caffeine or marijuana use.
- Smokers With Marijuana: People who smoke who have heavy marijuana use
- Total: Total of all reporting groups
Arm/Group | Non-smokers | Smokers Methol | Smokers Non Menthol | Smokers Without Comorbidities | Smokers With Caffeine | Smokers With Marijuana | Total
Number analyzed (Participants) | 47 | 22 | 41 | 34 | 22 | 18 | 184
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (13.4) | 43.1 (12.9) | 36.4 (14.2) | 39.1 (13.1) | 46.0 (12.9) | 42.3 (12.6) | 44 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 7 | 14 | 0 | 0 | 0 | 21
  Male | 47 | 15 | 27 | 34 | 22 | 18 | 163

OUTCOME MEASURES:

1. Primary Outcome: PET Scan, Rating Scales
Description: Vt/fp values (indicating relative densities of alpha4beta2 nicotinic acetylcholine receptors in different brain regions) in various brain regions - can also be referred to as mL/cm3.
Time Frame: Primary outcome measures will be determined over approximately 3 weeks
Population: Non-smokers and smokers (with the set of different conditions: menthol, non-menthol, w/ caffeine, w/ marijuana, w/o caffeine+marijuana) who underwent PET scanning to measure the total volume of distribution Vt in the prefrontal cortex.
Measure: Mean (Standard Deviation); unit: Vt/fp or mL/cm3
Groups:
- Smoker vs. Non Smoker: menthol smoker vs. non-menthol smoker vs. non smoker (w/o caffeine and marijuana) vs. smoker (w/o caffeine and marijuana) vs. smoker w/ caffeine use vs. smoker w/ marijuana use
Arm/Group | Smoker vs. Non Smoker
Number analyzed (Participants) | 184
Vt/fp or mL/cm3
  Non-smokers: number analyzed (Participants) | 47
  Non-smokers | 7.1 (1.3)
  Smokers menthol: number analyzed (Participants) | 22
  Smokers menthol | 8.6 (1.6)
  Smokers non-menthol: number analyzed (Participants) | 41
  Smokers non-menthol | 7.9 (1.2)
  Smokers w/o caff+marij: number analyzed (Participants) | 34
  Smokers w/o caff+marij | 8.0 (1.2)
  Smokers w/ caff: number analyzed (Participants) | 22
  Smokers w/ caff | 11.9 (5.7)
  Smokers w/ marij: number analyzed (Participants) | 18
  Smokers w/ marij | 10.8 (2.9)

ADVERSE EVENTS:
Time Frame: 3 weeks
Groups:
- Non-smokers: Participants who did not smoke.
- Smokers Methol: Participants who smoked menthol cigarettes.
- Smokers Non Menthol: Participants who smoked non menthol cigarettes
- Smokers Without Comorbidities: Participants who smoked without heavy use of caffeine or marijuana.
- Smokers With Caffeine: Participants who smoked with heavy caffeine use.
- Smokers With Marijuana: Participants who smoked with heavy marijuana use.
Arm/Group | Non-smokers | Smokers Methol | Smokers Non Menthol | Smokers Without Comorbidities | Smokers With Caffeine | Smokers With Marijuana
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/22 | 0/41 | 0/34 | 0/22 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/22 | 0/41 | 0/34 | 0/22 | 0/18
Other Adverse Events (participants affected / at risk) | 0/47 | 0/22 | 0/41 | 0/34 | 0/22 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No